CLINICAL TRIAL: NCT00904033
Title: A Pilot Study of the Effects of High-Dose Oral Calcitriol and Physical Activity on Bone Health in Breast Cancer Survivors
Brief Title: Calcitriol, Physical Activity, and Bone Health in Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Research Assistant Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RSRB00025478
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasms; Bone and Bones
MeSH Terms: conditions — Breast Neoplasms | interventions — Calcitriol; Exercise; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Multivitamin (Active Comparator): Multivitamin used as control group.
  Interventions: Dietary Supplement: Multivitamin
- Exercise (Experimental): Exercise consisting of progressive walking and resistance band training.
  Interventions: Behavioral: Exercise
- Calcitriol (Experimental): Calcitriol pill taken once per week.
  Interventions: Drug: Calcitriol
- Calcitriol and Exercise (Experimental): Calcitriol pill taken once per week plus Exercise consisting of progressive walking and resistance band training.
  Interventions: Drug: Calcitriol; Behavioral: Exercise

INTERVENTIONS:
Drug: Calcitriol — Calcitriol tablet taken once per week.
  Arms: Calcitriol; Calcitriol and Exercise
Behavioral: Exercise — Exercise consisting of progressive walking and resistance band training
  Arms: Calcitriol and Exercise; Exercise
Dietary Supplement: Multivitamin
  Other Names: Control
  Arms: Multivitamin

SUMMARY:
Both the calcitriol and exercise interventions are aimed at reducing fracture risk by maintaining proper bone density, thereby preventing osteoporotic/osteopenic conditions and increasing muscle mass. Both calcitriol and exercise are efficacious in maintaining proper bone health and muscle mass among the general population, but little research has been done on breast cancer patients and survivors. The combination of calcitriol and exercise, which function through different but similar mechanisms, could produce interactive effects in reducing fracture risk among breast cancer survivors.

Hypothesis: A combination of calcitriol along with a structured home-based walking and progressive resistance exercise program will be efficacious in preventing bone resorption and in increasing bone formation among survivors of invasive breast cancer.

DETAILED DESCRIPTION:
Primary Objective

To collect data on the efficacy and feasibility of a supplementation of calcitriol with/without an accompanying structured home-based walking/progressive resistance exercise program for improving bone health among breast cancer survivors.

Secondary Objectives

To collect data on the efficacy and feasibility of a supplementation of calcitriol with/without an accompanying structured home-based walking/progressive resistance exercise program for increasing strength among breast cancer survivors.

To collect data on the efficacy and feasibility of a supplementation of calcitriol with/without an accompanying structured home-based walking/progressive resistance exercise program for improving skeletal muscle mass among breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Must be female.
* Women of child-bearing potential (i.e. women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device (IUD), or double barrier device) and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Contraceptive use needs to be continued at least 1 month after the trial has ended.
* Must provide informed consent.
* Must be willing to discontinue use of calcium and/or vitamin D supplements.
* Participants must have an ionized serum calcium level within normal limits (1.19-1.29mmol/L) and a total corrected serum calcium of < 10.2mg/dl.
* Must have a functional capacity rating of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) performance status when assessed at baseline.
* Must have the approval of their treating physician (or physician's nurse practitioner or physician's assistant) to participate in sub-maximal physiological fitness testing and a low to moderate home-based walking and progressive resistance exercise program and to receive the 12-week supplementation of calcitriol 45 μg. Participants assigned to either of the calcitriol treatment arms will be instructed to stop taking calcium and/or vitamin D supplements.
* Must be less than five years from the diagnosis of breast cancer and have received chemotherapy, radiation therapy, and/or hormonal therapy. Chemotherapy and radiation therapy, if received, must have been completed prior to study enrollment. Hormonal therapy may be ongoing.

Exclusion Criteria:

* Subjects with life-threatening conditions that would preclude them from breast cancer treatment including chronic cardiac failure, which is unstable despite medication use, uncontrolled hypertension, uncontrolled diabetes mellitus, or unstable coronary artery disease.
* Patients who had a myocardial infarction within the past year.
* Patients with severe metabolic disorders, which includes phenylketonuria (PKU), homocystinuria, and Fabry's disease, that would preclude them from taking calcitriol.
* Patients with impaired renal function (CRCL < 60 mL/min) or who had kidney stones (calcium salt) within the past 5 years.
* Patients with hypercalcemia (corrected serum Ca > 10.2 mg/dl) or a history of hypercalcemia or vitamin D toxicity.
* Patients currently taking calcium supplements or aluminum-based antacids must be willing to discontinue their use if they are to enroll in the study.
* Patients currently taking vitamin D supplements must immediately discontinue their use if they are to enroll in the study.
* Patients with a known sensitivity to calcitriol.
* Women who are pregnant or lactating.
* Previously verified diagnosed of osteoporosis.
* Women on antiresorptive drugs (e.g. bisphosphonates) within the past year.
* Patients not capable of participating in an exercise intervention due to severe knee arthrosis or ligament/cartilage injuries of the lower extremities.
* Women currently using oral contraception.
* Women with malabsorptive syndromes (i.e. cystic fibrosis, chronic pancreatitis) or taking medications that decrease the absorption of fat soluble vitamins (i.e. Orlistat, Questran).
* Participants assigned to calcitriol who are routinely taking a multivitamin supplement may continue the supplement as long as the amount of vitamin D in the supplement is not in excess of the RDA (recommended daily allowance) of 400 IU or 10 μg. If they are not taking a multivitamin supplement, they will be asked to not start supplementation while on study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke J Peppone, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Multivitamin: Multivitamin used as control group.
  Multivitamin
- Exericse: Exercise consisting of progressive walking and resistance band training.
  Exercise: Exercise consisting of progressive walking and resistance band training
Period: Overall Study
Arm/Group | Multivitamin | Exericse | Calcitriol | Calcitriol and Exercise
Started | 10 | 10 | 10 | 11
Completed | 9 | 9 | 9 | 9
Not Completed | 1 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Unable to obtain final blood draw | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multivitamin | Exericse | Calcitriol | Calcitriol and Exercise | Total
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (8.2) | 55.8 (6.7) | 52.0 (6.8) | 55.1 (8.7) | 53.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 11 | 41
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 10 | 8 | 11 | 38
  Not White | 1 | 0 | 2 | 0 | 3
Marital Status [Count of Participants; unit: Participants]
  Married | 6 | 7 | 9 | 11 | 33
  Single/Divorced/Widowed | 4 | 3 | 1 | 0 | 8
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 6 | 1 | 5 | 3 | 15
  Postmenopausal | 4 | 9 | 5 | 8 | 26
Hormonal Therapy [Count of Participants; unit: Participants] — Population: Subject did not received hormone therapy.
  Participants
    number analyzed (Participants) | 10 | 9 | 10 | 11 | 40
    Tamoxifen | 7 | 4 | 6 | 4 | 21
    Aromatase Inhibitor | 3 | 5 | 4 | 7 | 19
Stage of Cancer [Count of Participants; unit: Participants] — Stage 0. This stage describes cancer in situ, which means "in place." Stage 0 cancers are located in the place they started and have not spread to nearby tissues.
  Stage I. This stage is usually a small cancer that has not grown deeply into nearby tissues.
  Stage II and Stage III. In general, these 2 stages indicate larger cancers that have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not to other parts of the body.
  Stage IV. This stage means that the cancer has spread to other organs or parts of the body.
  Stage 0 is best, Stage IV is worst.
  Participants
    0 / I | 3 | 2 | 5 | 7 | 17
    II | 4 | 6 | 4 | 3 | 17
    III | 3 | 2 | 1 | 1 | 7
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 7 | 7 | 7 | 6 | 27
  No | 3 | 3 | 3 | 5 | 14
Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 10 | 10 | 10 | 11 | 41
  No | 0 | 0 | 0 | 0 | 0
Current Cardiovascular Exercise [Count of Participants; unit: Participants]
  Yes | 5 | 6 | 6 | 7 | 24
  No | 5 | 4 | 4 | 4 | 17
Current Resistance Training [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2 | 3 | 7
  No | 8 | 10 | 8 | 8 | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Measure Description: Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Values below 18.5 represent "Underweight", 18.5 to 24.9 represent "Normal or Healthy Weight", 25.0 to 29.9 represent "Overweight" and 30.0 and above represent "Obese". Population: There were 5 subjects who did not have a body weight available (4 subjects in the multivitamin arm and 1 subject in the Calcitriol and Exercise arm) and therefore a BMI was not possible to calculate.
  kg/m^2
    number analyzed (Participants) | 6 | 10 | 10 | 10 | 36
    (all) | 31.3 (6.0) | 32.4 (7.5) | 28.4 (5.5) | 28.1 (3.6) | 29.9 (5.9)
Serum NTx - Bone Resorption [Mean (Standard Deviation); unit: nm BCE] — Serum NTx level is used to aid in predicting skeletal response (bone mineral density) to antiresorptive therapy and in monitoring bone resorption changes following initiation of antiresorptive therapy. The measurement range is in nanoMoles (nm) Bone Collagen Equivalents (BCE). Population: Serum NTx not recorded for two subjects in the Calcitriol and Exercise arm because their values were out of range and were not used per the instructions of the assay kit used for Serum NTx analysis.
  nm BCE
    number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
    (all) | 12.2 (10.0) | 11.6 (5.7) | 13.4 (8.1) | 14.4 (9.5) | 12.9 (8.2)
Serum BSAP - Bone Formation [Mean (Standard Deviation); unit: ng/ml] — The Bone-Specific Alkaline Phosphatase (BSAP) assay provides a general index of bone formation and a specific index of total osteoblast activity. BSAP and osteocalcin are the most effective markers of bone formation and are particularly useful for monitoring bone formation therapies and antiresorptive therapies. Population: Serum BSAP not recorded for 1 subject in the Calcitriol and Exercise arm because the values were out of range and were not used per the instructions of the Serum BSAP assay kit.
  ng/ml
    number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
    (all) | 12.2 (7.1) | 13.8 (7.2) | 12.2 (7.4) | 12.0 (5.6) | 12.6 (6.7)
Serum BMOI - Bone Metabolism Index [Mean (Standard Deviation); unit: Z-Score] — BMOI is defined as follows:
  ΔZ BSAP - ΔZ NTx, where ZBSAP = (BSAPObserved-BSAPμ at baseline)/σ (standard deviation) at baseline, and ZNTx = (NTxObserved-NTxμ at baseline)/σ at baseline. A positive number for the BMOI indicates a net bone gain: i.e., resorption decreased and formation increased over the course of the intervention. A negative number for the BMOI indicates net bone loss: i.e., resorption increased and formation decreased over the course of the intervention. Population: Serum BMOI not recorded for two subjects in the Calcitriol and Exercise arm because their values were out of range and were not used per the instructions of the Serum BMOI assay kit.
  Z-Score
    number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
    (all) | 0.03 (1.25) | 0.34 (1.05) | -0.12 (1.44) | -0.26 (0.96) | 0.01 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Bone Resorption (Exercise)
Description: Bone Resorption using Serum NTx (Exercise comparison)
  Serum NTx level is used to aid in predicting skeletal response (bone mineral density) to antiresorptive therapy and in monitoring bone resorption changes following initiation of antiresorptive therapy. Elevated levels of serum NTx indicate elevated bone resorption. Elevated bone resorption is the primary cause of agerelated bone loss and that low bone mass often results in osteopenia and is the major cause of osteoporosis. The measurement range is in nanoMoles (NM) Bone Collagen Equivalents (BCE).
Time Frame: Week 12
Population: No Exercise group consists of Multivitamin and Calcitriol arms N=20; Exercise group consists of Exercise and Calcitriol+Exercise arms N=19**
  ** 2 subjects have missing data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: nm BCE
Groups:
- No Exercise: Multivitamin Arm + Calcitriol Arm:Calcitriol pill taken once per week
- Exercise: Exercise Arm: Exercise consisting of progressive walking and resistance band training
  Calcitriol+ Exercise Arm: Calcitriol pill taken once per week + Exercise
Arm/Group | No Exercise | Exercise
Number analyzed (Participants) | 20 | 19
nm BCE | 13.8 (1.656) | 14.7 (1.033)
Statistical Analysis 1: Comparison: No Exercise vs Exercise; Test type: Other; p = 0.86, ANCOVA; Main Effects Results only for No Exercise vs Exercise

2. Primary Outcome: Bone Resorption (Calcitriol)
Description: Bone Resorption using Serum NTx (Calcitriol comparison)
  Serum NTx level is used to aid in predicting skeletal response (bone mineral density) to antiresorptive therapy and in monitoring bone resorption changes following initiation of antiresorptive therapy. Elevated levels of serum NTx indicate elevated bone resorption. Elevated bone resorption is the primary cause of agerelated bone loss and that low bone mass often results in osteopenia and is the major cause of osteoporosis. The measurement range is in nanoMoles (nm) Bone Collagen Equivalents (BCE).
Time Frame: Week 12
Population: No Calcitriol group consists of Multivitamin arm and Exercise arm N=20; Calcitriol group consists of Calcitriol and Calcitriol+Exercise arms N=19**
  ** 2 subjects have missing data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: nm BCE
Groups:
- No Calcitriol: Multivitamin Arm + Exercise Arm:Exercise consisting of progressive walking and resistance band training
- Calcitriol: Calcitriol Arm: Calcitriol pill taken once per week
  and
  Calcitriol+Exercise Arm:Exercise consisting of progressive walking and resistance band training
Arm/Group | No Calcitriol | Calcitriol
Number analyzed (Participants) | 20 | 19
nm BCE | 12.5 (1.785) | 15.0 (1.113)
Statistical Analysis 1: Comparison: No Calcitriol vs Calcitriol; Test type: Other; p = 0.19, ANCOVA

3. Primary Outcome: Bone Formation (Exercise)
Description: Bone Formation using Serum BSAP (Exercise comparison)
  The Bone-Specific Alkaline Phosphatase (BSAP) assay provides a general index of bone formation and a specific index of total osteoblast activity. BSAP and osteocalcin are the most effective markers of bone formation and are particularly useful for monitoring bone formation therapies and antiresorptive therapies.
Time Frame: Week 12
Population: No Exercise group consists of Multivitamin and Calcitriol arms N=20; Exercise group consists of Exercise and Calcitriol+Exercise arms N=20**
  **1 subject has missing data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | No Exercise | Exercise
Number analyzed (Participants) | 20 | 20
ng/ml | 13.8 (1.513) | 14.7 (0.957)
Statistical Analysis 1: Comparison: No Exercise vs Exercise; Test type: Other; p = 0.49, ANCOVA

4. Primary Outcome: Bone Formation (Calcitriol)
Description: Bone Formation using Serum BSAP (Calcitriol comparison)
  The Bone-Specific Alkaline Phosphatase (BSAP) assay provides a general index of bone formation and a specific index of total osteoblast activity. BSAP and osteocalcin are the most effective markers of bone formation and are particularly useful for monitoring bone formation therapies and antiresorptive therapies.
Time Frame: Week 12
Population: No Calcitriol group consists of Multivitamin arm and Exercise arm N=20; Calcitriol group consists of Calcitriol and Calcitriol+Exercise arms N=20**
  ** 1 subject has missing data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Groups:
- Calcitriol: Calcitriol Arm: Calcitriol pill taken once per week
  and
  Calcitriol+ Exercise Arm:Exercise consisting of progressive walking and resistance band training
Arm/Group | No Calcitriol | Calcitriol
Number analyzed (Participants) | 20 | 20
ng/ml | 12.0 (1.268) | 16.3 (0.802)
Statistical Analysis 1: Comparison: No Calcitriol vs Calcitriol; Test type: Other; p < 0.01, ANCOVA

5. Secondary Outcome: Handgrip (kg) Strength - (Exercise)
Description: Handgrip (kg) Strength (Exercise comparison)
  Hand grip strength can be quantified by measuring the amount of static force that the hand can squeeze around a dynamometer. It is typically measured in kilograms or pounds and varies by sex and age. Normative data for females is AGE 35-39 --> 20.3-34.1kg; AGE 40-44 --> 18.9-32.7kg; AGE 45-49 --> 18.6-32.4kg; AGE 50-54 --> 18.1-31.9kg; AGE 55-59 --> 17.7-31.5kg; AGE 60-64 --> 17.2-31.0kg; AGE 65-69 --> 15.4-27.2kg; AGE 70-99 --> 14.7-24.5kg. Values less than the normal range are considered weak strength. Values greater than the normal range are considered strong strength.
Time Frame: Week 12
Population: No Exercise group consists of Multivitamin and Calcitriol arms N=14*; Exercise group consists of Exercise and Calcitriol+Exercise arms N=17** * 6 subjects have missing data for this outcome.
  ** 4 subjects have missing data for this outcome.
Measure: Mean (Standard Error); unit: kg
Arm/Group | No Exercise | Exercise
Number analyzed (Participants) | 14 | 17
kg | 26.6 (1.633) | 27.8 (0.919)
Statistical Analysis 1: Comparison: No Exercise vs Exercise; Test type: Other; p = 0.16, t-test, 2 sided

6. Secondary Outcome: Handgrip (kg) Strength - (Calcitriol)
Description: Handgrip (kg) Strength - (Calcitriol comparison)
  Hand grip strength can be quantified by measuring the amount of static force that the hand can squeeze around a dynamometer. It is typically measured in kilograms or pounds and varies by sex and age. Normative data for females is AGE 35-39 --> 20.3-34.1kg; AGE 40-44 --> 18.9-32.7kg; AGE 45-49 --> 18.6-32.4kg; AGE 50-54 --> 18.1-31.9kg; AGE 55-59 --> 17.7-31.5kg; AGE 60-64 --> 17.2-31.0kg; AGE 65-69 --> 15.4-27.2kg; AGE 70-99 --> 14.7-24.5kg. Values less than the normal range are considered weak strength. Values greater than the normal range are considered strong strength.
Time Frame: Week 12
Population: No Calcitriol group consists of Multivitamin arm and Exercise arm N=14*; Calcitriol group consists of Calcitriol and Calcitriol+Exercise arms N=17** * 6 subjects have missing data for this outcome.
  ** 4 subjects have missing data for this outcome.
Measure: Mean (Standard Error); unit: kg
Arm/Group | No Calcitriol | Calcitriol
Number analyzed (Participants) | 14 | 17
kg | 27.4 (1.441) | 27.1 (0.804)
Statistical Analysis 1: Comparison: No Calcitriol vs Calcitriol; Test type: Other; p = 0.84, t-test, 2 sided

7. Secondary Outcome: Body Mass Index (Exercise)
Description: Body Mass Index (BMI) - (Exercise Comparison)
  Measure Description: Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Values below 18.5 represent "Underweight", 18.5 to 24.9 represent "Normal or Healthy Weight", 25.0 to 29.9 represent "Overweight" and 30.0 and above represent "Obese".
Time Frame: Week 12
Population: No Exercise group consists of Multivitamin and Calcitriol arms N=16*; Exercise group consists of Exercise and Calcitriol+Exercise arms N=20** *4 subjects have missing data for this outcome.
  **1 subject has missing data for this outcome.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | No Exercise | Exercise
Number analyzed (Participants) | 16 | 20
kg/m^2 | 30.0 (0.312) | 30.2 (0.185)
Statistical Analysis 1: Comparison: No Exercise vs Exercise; Test type: Other; p = 0.38, t-test, 2 sided

8. Secondary Outcome: Body Mass Index (Calcitriol)
Description: Body Mass Index(BMI) - (Calcitriol comparison)
  Measure Description: Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Values below 18.5 represent "Underweight", 18.5 to 24.9 represent "Normal or Healthy Weight", 25.0 to 29.9 represent "Overweight" and 30.0 and above represent "Obese".
Time Frame: Week 12
Population: No Calcitriol group consists of Multivitamin arm and Exercise arm N=16*; Calcitriol group consists of Calcitriol and Calcitriol+Exercise arms N=20** * 4 subjects have missing data for this outcome.
  ** 1 subject has missing data for this outcome.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | No Calcitriol | Calcitriol
Number analyzed (Participants) | 16 | 20
kg/m^2 | 30.1 (0.284) | 30.1 (0.161)
Statistical Analysis 1: Comparison: No Calcitriol vs Calcitriol; Test type: Other; p = 0.92, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Multivitamin | Exericse | Calcitriol | Calcitriol and Exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 6/10 | 6/10 | 5/10 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multivitamin (N=10) | Exericse (N=10) | Calcitriol (N=10) | Calcitriol and Exercise (N=11)
Hypercalcemia - Grade 1 (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Creatinine Elevation - Grade 1 (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0
Hyperkalemia - Grade 1 (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Hypernatremia - Grade 1 (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypergycemia - Grade 1 (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1
Hyperglycemia - Grade 2 (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood Urea Nitrogen Elevation - Grade 1 (Blood and lymphatic system disorders) | 3 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-05-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT00904033/Prot_SAP_000.pdf